CLINICAL TRIAL: NCT02297100
Title: The Impact of Injection Location on the Efficacy of Intravesicular Onabotulinumtoxin A in Interstitial Cystitis--Phase 4
Brief Title: Intravesicular Onabotulinumtoxin A in Interstitial Cystitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00026734
Record Dates: First submitted 2014-09-30; First posted 2014-11-21 (Estimated); Results first posted 2018-05-22 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Interstitial Cystitis
Keywords: women; interstitial cystitis; bladder pain syndrome; botox; onabotulinum toxin A
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Botox upper aspect trigone (Experimental): Subjects in the experimental cohort will receive a one time dose of 100 units of Onabotulinumtoxin A diluted in 10 mL of preservative free normal saline and injected in 1.0 mL boluses in a set pattern across the upper aspect of the trigone of the urinary bladder.
  Interventions: Drug: Onabotulinumtoxin A; Procedure: injections upper aspect of trigone of urinary bladder
- botox periphery of trigone (Active Comparator): Each group will receive a total of 100 units of botox spread out among 10 separate injections. Subjects in the control group will have 10 injections made about the periphery of the trigone. The control cohort will receive a one time dose of Onabotulinumtoxin A using the same dilution and number of boluses, but boluses will be administered at random sites on the posterior bladder wall (excluding the trigone).
  Interventions: Drug: Onabotulinumtoxin A; Procedure: injections on posterior bladder wall excluding the trigone

INTERVENTIONS:
Drug: Onabotulinumtoxin A — 100 units of botox spread out among 10 separate injections
  Other Names: Botox
Procedure: injections upper aspect of trigone of urinary bladder — We hypothesize that injections into the trigone should be more effective in the treatment of IC than injections elsewhere in the bladder.
  Arms: Botox upper aspect trigone
Procedure: injections on posterior bladder wall excluding the trigone — We hypothesize that injections into the trigone should be more effective in the treatment of IC than injections elsewhere in the bladder.
  Arms: botox periphery of trigone

SUMMARY:
The purpose of this research study is to identify the optimal usage of Onabotulinumtoxin A in interstitial cystitis. Onabotulinumtoxin A, more commonly known by the trade name Botox®, is a medication that comes from the bacteria Clostridium botulinum. It works by blocking the release of the neurotransmitter acetylcholine(a chemical messenger that carries signals between nerve cells and other cells in the body). Blocking that neurotransmitter results in decreased muscle activity.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy of intravesicular Onabotulinumtoxin A injections for the treatment of interstitial cystitis (IC). Specifically, we hypothesize that trigonal Onabotulinumtoxin A injections is an effective treatment for IC and will result in more subjective and objective symptom relief than posterior wall Onabotulinumtoxin A injections.

ELIGIBILITY:
Inclusion Criteria:

1. Adult females between the ages of 18 and 80 inclusive
2. Patients being treated for IC who are refractory to conservative management and oral therapy.
3. willing and able to initiate catheterization post-treatment

Exclusion Criteria:

1. Any history of bladder cancer, uterine cancer, ovarian cancer, vaginal cancer, urethral diverticulum, spinal cord injury, stroke, Parkinson's disease, multiple sclerosis, spina bifida, cyclophosphamide treatment, radiation treatment to the pelvis, bladder tuberculosis, genital herpes.
2. Currently on or requiring anti-platelet/anti-coagulant concomitant therapy or having been on anti-platelet/ anti-coagulant therapy within the past 3 months
3. Pregnancy. Pregnancy is an absolute contraindication to undergoing these procedures. Thus, as part of their normal pre-operative work up, which is standard of care, pregnancy tests are administered if they are women of child-bearing age, are sexually active, and are within 10 days of the normal menstrual period. If positive, they will be excluded as they will not undergo the procedure.
4. An active urinary tract infection as shown during clean-catch urinalysis at screening visit. Subject may be re-screened if UTI is successfully treated and urinalysis is negative at rescreening.
5. A history of hypersensitivity or allergy to any botulinum toxin preparation
6. A post-void residual (PVR) urine volume >200mL at baseline
7. Treatment with botulinum toxin during the 12 week period prior to the trial

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Evans, M.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botox Upper Aspect Trigone | Botox Periphery of Trigone
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botox Upper Aspect Trigone | Botox Periphery of Trigone | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.38 (13.64) | 46.5 (12.32) | 47.41 (12.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 13 | 13 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 12 | 13 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Will be Assessing the Measurement of Subjective Patient Pain Using the O'Leary-Sant Symptom and Problem Indexes.
Description: The O'Leary-Sant is one questionnaire that assesses the severity of symptoms and the how much of a problem the symptoms cause for the patient and it provides two scores. The scores ranges for the symptoms is 0-20 and for how bothersome the symptoms are, the score range is 0-16. Higher scores for both denotes worse outcomes.
Time Frame: 30 and 90 days post treatment
Population: One participant was lost to follow-up in the experimental group and no data was collected at 30 days on one participant in the control group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botox Upper Aspect Trigone | Botox Periphery of Trigone
Number analyzed (Participants) | 12 | 14
units on a scale
  Symptoms @ 30 days: number analyzed (Participants) | 12 | 13
  Symptoms @ 30 days | 10.92 (3.15) | 10.85 (4.18)
  Bother @ 30 days: number analyzed (Participants) | 12 | 13
  Bother @ 30 days | 9.75 (4.00) | 9.92 (4.61)
  Symptoms @ 90 days | 10.75 (3.62) | 12.00 (4.54)
  Bother @ 90 days | 10.17 (3.16) | 10.29 (4.07)

2. Primary Outcome: The Primary Outcome Will be Assessing the Measurement of Subjective Patient Pain Using the Pelvic Pain and Urinary Urgency Frequency (PUF) Questionnaire
Description: The PUF questionnaire evaluates symptoms of pain and how much they bother the patient. Two score are given and added together to produce a total score. The score range for symptoms is 0-28 and the range for bother is 0-16. Higher scores denotes worse outcomes.
Time Frame: 30 and 90 days post-treatment
Population: One participant from the experimental group was lost to follow-up. Data was not collected at 30 days for bother and symptom for one participant in the control group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botox Upper Aspect Trigone | Botox Periphery of Trigone
Number analyzed (Participants) | 12 | 14
units on a scale
  Symptoms @ 30 days: number analyzed (Participants) | 12 | 13
  Symptoms @ 30 days | 13.83 (4.90) | 12.31 (4.71)
  Bother @ 30 days: number analyzed (Participants) | 12 | 13
  Bother @ 30 days | 7.33 (2.77) | 7.31 (3.17)
  Symptoms @ 90 days | 13.33 (4.75) | 13.21 (4.42)
  Bother @ 90 days | 7.25 (2.83) | 7.5 (2.77)

3. Secondary Outcome: Change in Patient Performance in Uroflowmetry.
Description: Uroflowmetry is a test that measures the volume of urine released from the body, the speed with which it is released, and how long the release takes.
Time Frame: 30 days and 90 days post treatment
Population: No data was collected for two participants in the experimental group and one participant in the control group at 30 days. No data was collected for one participant in the experimental group at 90 days.
Measure: Mean (Standard Deviation); unit: ml/s
Arm/Group | Botox Upper Aspect Trigone | Botox Periphery of Trigone
Number analyzed (Participants) | 12 | 14
ml/s
  @ 30 days: number analyzed (Participants) | 11 | 13
  @ 30 days | 11.82 (5.64) | 9.5 (7.83)
  @ 90 days | 12.17 (7366) | 15.5 (11.89)

4. Other Pre Specified Outcome: Secondary Outcomes Will be Assessing Change in Patient Performance in Post Void Residuals.
Time Frame: 30 days and 90 days post treatment
Population: Data was not collected on one participant in the experimental group at 30 and 90 days post treatment. Data was not collected on two individuals at 30 days post treatment in the control group.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Botox Upper Aspect Trigone | Botox Periphery of Trigone
Number analyzed (Participants) | 12 | 14
mL
  @ 30 days: number analyzed (Participants) | 12 | 12
  @ 30 days | 27.17 (37.06) | 35.33 (48.00)
  @ 90 days | 38.92 (48.10) | 60.64 (71.38)

ADVERSE EVENTS:
Time Frame: baseline, up to 4 years
Arm/Group | Botox Upper Aspect Trigone | Botox Periphery of Trigone
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 4/13 | 7/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Botox Upper Aspect Trigone (N=13) | Botox Periphery of Trigone (N=14)
Painful Voiding (Renal and urinary disorders) | 0 | 1
Urethral Edema (Renal and urinary disorders) | 1 | 0
Urgency (Renal and urinary disorders) | 1 | 2
Urinary Tract Infection (Renal and urinary disorders) | 2 | 2
Retention (Renal and urinary disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT02297100/Prot_SAP_000.pdf